CLINICAL TRIAL: NCT00118612
Title: A DoubleBlind Phase 2b Study to Evaluate Safety & Efficacy of Different Doses of Tyrosine Adsorbed Birch+Hazel+Alder Pollen Allergoid With MPL® in Patients Sensitized to Birch, Hazel, Alder Pollen
Brief Title: Different Doses of Tyrosine Adsorbed Tree Pollen Allergoid With Monophosphoryl Lipid A (MPL) in Patients Sensitized to Tree Pollen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TreeMATAMPL203; P2DP05003
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Specific Immunotherapy; Allergy Vaccination; Allergenicity
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes

ARMS (4):
- Therapeutic Regimen (Experimental)
  Interventions: Biological: Tree MATA MPL - Therapeutic Regimen
- Intermediate dose (Experimental)
  Interventions: Biological: Tree MATA MPL - Intermediate dose
- Low dose (Experimental)
  Interventions: Biological: Tree MATA MPL - Low dose
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tree MATA MPL - Therapeutic Regimen — 600, 1600, 4000, 4000 SU/0.5 mL
  Arms: Therapeutic Regimen
Biological: Tree MATA MPL - Intermediate dose — 300, 600, 1600, 1600 SU/0.5 mL
  Arms: Intermediate dose
Biological: Tree MATA MPL - Low dose — 300, 300, 300, 300 SU/0.5 mL
  Arms: Low dose
Biological: Placebo — L-tyrosine 2% w/v , 4 injections
  Arms: Placebo

SUMMARY:
Allergen-specific immunotherapy (SIT), the administration of gradually increasing quantities of an allergen extract to an allergic patient, is a curative approach which directly treats the underlying allergic disease. Tree MATA MPL has been developed to provide pre-seasonal specific immunotherapy for patients with an allergy to tree pollen (hay fever).

The purpose of this double-blind Phase IIb study is to assess the tolerability and immunogenicity of different doses of Tree MATA MPL in volunteers allergic to birch, hazel and alder pollen.

DETAILED DESCRIPTION:
Tree MATAMPL (tyrosine adsorbed tree pollen allergoid with monophosphoryl lipid A (MPL®)) has been developed to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to cross-reacting tree pollens that cause rhinitis and/or conjunctivitis with or without mild to moderate asthma.

This was a phase IIb, double-blind, placebo-controlled study to assess the tolerability and immunogenicity of different doses of Tree MATA MPL in volunteers allergic to birch, hazel and alder pollen.

Sixty eight (68) volunteers were randomly assigned to one of three active treatments or placebo to receive up to 4 subcutaneous injections of either increasing doses of Tree MATAMPL or Placebo over 7 day (+1 day) interval.

The duration of the study from screening (Visit 1) to end of study (Visit 6, Post-Treatment Visit) was approximately 50 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a positive skin prick test for birch and hazel and alder allergen.
* Positive skin prick test to positive histamine control
* Negative skin prick test to negative control
* Specific IgE for birch as documented by radioallergosorbent or equivalent test with class ≥ 2
* History of at least 1 season of moderate to severe seasonal rhinoconjunctivitis due to an IgE - mediated allergy to pollen from birch, hazel, and alder
* Patients must score on the disease severity questionnaire as moderate or severe.
* Males or non-pregnant, non-lactating females
* Patients who are normally active and otherwise judged to be in good health
* Patients must be willing and able to attend required study visits.
* Patients must be able to follow instructions.
* Patients must be willing and able to give written informed consent and must provide this consent.

Exclusion Criteria:

* Acute or subacute atopic dermatitis and/or urticaria factitia and/or urticaria due to physical or chemical influence and/or chronic dermatitis
* Moderate to severe asthma
* Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the skin prick test; both forearms must be available for testing.
* History or presence of diabetes, cancer or any clinically significant cardiac, metabolic, renal, or hematologic diseases or disorders
* Recent clinically significant history of hepatic, gastrointestinal, dermatologic, venereal, neurologic or psychiatric diseases or disorders
* Any clinically significant abnormal laboratory value at Visit 1
* Perennial allergens: clinically relevant sensitivity to house dust mites, molds, and epithelia
* Patient has clinically relevant sensitivity to the following summer/autumn season flowering plants: plantain, orache, nettle, mugwort, Parietaria judaica, Bermuda grass, or ragweed.
* Secondary alteration at the affected organ
* History of autoimmune diseases and/or rheumatoid diseases
* Patient is taking ß-blockers for any indication including eye drops
* Patient who is not allowed to receive adrenalin
* Patients in whom tyrosine metabolism is disturbed
* Presence of a disease with a pathogenesis interfering with the immune response and patient has received medication which could influence the results of this study
* Acute or significant chronic infection
* History of anaphylaxis
* Documented history of angioedema
* Hypersensitivity to excipients in the study medications
* Previous or current immunotherapy with comparable tree allergen extracts
* Currently using anti-allergy medication and other drugs with antihistaminic activity
* Patients currently participating in a clinical trial or who have been exposed to study medication within the last 30 days
* Patients who cannot communicate reliably with the Investigator or who are not likely to cooperate with the requirements of the study
* Patient is pregnant or planning pregnancy and/or lactating
* Patient has received treatment with preparation containing MPL during the past 12 months
* Concurrent use of any prohibited medication(s), as listed in the study protocol, or inadequate washout of any medication
* Any systemic disorder that could interfere with the evaluation of the study medication(s)
* Clinical history of drug or alcohol abuse, at the Investigator's discretion, that would interfere with the patient's participation in the study
* Study site staff or immediate relatives of study site staff or other individuals who would have access to the clinical study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2005-07-07 (Actual); Primary Completion 2005-09-15 (Actual); Study Completion 2005-09-15 (Actual)

PRIMARY OUTCOMES:
Immunological response to the three Tree MATA MPL treatment arms compared to placebo (birch specific) | Up to two approximately 2 months
  Efficacy was assessed based on the immunological differences between the three Tree MATA MPL treatment arms compared to placebo with respect to immunoglobulins (specific IgG, specific IgG1, specific IgG4, and specific IgE) for birch, alder, and hazel.

SECONDARY OUTCOMES:
Tolerability of individual subcutaneous doses | Up to two approximately 2 months
Tolerability of the cumulative subcutaneous doses | Up to two approximately 2 months
safety laboratory evaluation - clinical chemistry | Up to two approximately 2 months
safety laboratory evaluation - hematology | Up to two approximately 2 months
safety laboratory evaluation - urinalysis | Up to two approximately 2 months
Vital signs | Up to two approximately 2 months
Physical examinations | Up to two approximately 2 months
  Abnormal physical examination findings were summarized by clinical significance(CS or NCS) using frequencies and percentages of patients for each body system and overall
12-Lead ECGs | Up to two approximately 2 months
  QRS duration, PR interval, QT interval, and QTc
number of adverse events | Approximately 2 months
number of adverse reactions | Up to two approximately 2 months
immunological response to the three Tree MATA MPL treatment arms compared to placebo (alder and hazel specific) | Up to two approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Allied Research International Inc.
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada